CLINICAL TRIAL: NCT06060002
Title: Role of Prophylactic Biliary Stent in Reducing the Recurrence of Choledocholithiasis and Biliary Complications After Stone Clearance in Patients Awaiting Cholecystectomy-A Multicentric Randomized Controlled Trial (STONE Trial)
Brief Title: Role of Prophylactic Biliary Stent in Reducing the Recurrence of Choledocholithiasis
Acronym: STONE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: STONE_1
Record Dates: First submitted 2023-09-13; First posted 2023-09-29 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Patients will undergo stent removal and cholangiogram at 3 months of follow up (Active Comparator): In group A, patients will undergo stent removal and cholangiogram at 3 months of follow up. If we detect recurrent stone/s on cholangiogram, clearance will be done accordingly. If the patient is dated for cholecystectomy beyond 3 months then stent exchange will be done and patient will be followed up till they undergo cholecystectomy. During this waiting period in the later group, patients will undergo monthly follow up for development of any new onset symptoms that are suggestive of biliary pain, pancreatitis, cholangitis and cholecystitis.
  Interventions: Procedure: Group A - Stent exchange if cholecystectomy dated beyond 3 months
- Group B - Patients will undergo endoscopic ultrasound (EUS) at 3 months of follow up. (Sham Comparator): In group B, patients will undergo endoscopic ultrasound (EUS) at 3 months of follow up. If we detect recurrent stone/s in EUS then ERC and clearance will be done accordingly. Those who are dated for cholecystectomy beyond 3 months will undergo monthly follow up clinically (biliary pain, pancreatitis, cholangitis and cholecystitis) till they undergo cholecystectomy.
  Those patient in group B who are unwilling for EUS will be requested to get an magnetic resonance cholangiopancreatography (MRCP) while those unwilling for both EUS/MRCP will be followed up with ultrasound abdomen and liver function test (LFT).
  Interventions: Diagnostic Test: Group B - Diagnostic EUS/MRCP/USG abdomen and LFT at 3 months

INTERVENTIONS:
Procedure: Group A - Stent exchange if cholecystectomy dated beyond 3 months — Stent removal and cholangiogram and stone clearance (if recurrent stone/s is/are found). Stent exchange if cholecystectomy dated beyond 3 months
  Arms: Group A - Patients will undergo stent removal and cholangiogram at 3 months of follow up
Diagnostic Test: Group B - Diagnostic EUS/MRCP/USG abdomen and LFT at 3 months — Diagnostic EUS/MRCP/USG abdomen and LFT at 3 months to see recurrence of CDL. ERC and stone clearance (if recurrent stone/s found on EUS/MRCP/USG abdomen)
  Arms: Group B - Patients will undergo endoscopic ultrasound (EUS) at 3 months of follow up.

SUMMARY:
We planned this multicenter randomized controlled trial to study the role of a prophylactic biliary stent in recurrence of stones and biliary complications in patients awaiting cholecystectomy after biliary stone clearance

DETAILED DESCRIPTION:
Patients with cholelithiasis can have presence of concomitant choledocholithiasis (CDL) in upto 30%. These stones may remain asymptomatic or cause obstructive jaundice and complications like cholangitis and pancreatitis. In situations where there is a failure of CDL clearance during endoscopic retrograde cholangiography (ERC), biliary stenting is recommended to prevent complications. However, the role of prophylactic biliary stenting in situations where CDL clearance has been achieved, and the patient is awaiting cholecystectomy is debatable. One retrospective study showed benefit while a small prospective study and a retrospective study did not show benefit of prophylactic biliary stenting. Moreover, a randomized controlled trial addressing this question is lacking. Hence, we planned this multicenter randomized controlled trial to study the role of a prophylactic biliary stent in recurrence of stones and biliary complications in patients awaiting cholecystectomy after biliary stone clearance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-80 years
* Cases of cholelithiasis with concomitant CDL in whom CBD clearance is achieved will be included.

Exclusion Criteria:

* Informed consent not available
* Patients opting for single stage surgery
* Previous hepatobiliary surgery
* Failure to completely clear CDL on ERC
* Concomitant benign biliary strictures (like chronic pancreatitis, portal cavernoma cholangiopathy, post cholecystectomy, primary biliary cholangitis related)
* Previous cholecystectomy patients
* Associated malignancy
* Coagulopathy(INR>1.5, platlets<1lac)
* Severe cholangitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
To compare the CDL recurrence rate between the 2 groups | 3 Months

SECONDARY OUTCOMES:
To compare the pancreatic complications between the 2 groups -To compare the need for repeat ERC between the 2 groups The outcomes will be compared during the time period of 3 months irrespective of the timing of cholecystectomy. | 3 Months
To compare the biliary complications between the 2 groups | 3 Months